CLINICAL TRIAL: NCT07373067
Title: A Phase 1b Extension Trial To Allow Repeat Intracerebroventricular Injections of Ex Vivo Expanded, Autologous Adipose-Derived Stem Cells (RB-ADSCs) in Subjects Previously Treated in RBI Protocol RB-ADSC-02
Brief Title: Repeat Intracerebroventricular Injections of RB-ADSC in Subjects Previously Treated in RBI Protocol RB-ADSC-02
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneration Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-ADSC-02E
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: AD; Autologous; Stem cells; Cell therapy; Alzheimer Disease; RB-ADSC
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RB-ADSC low dose (Experimental): Participants will receive 2x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir every 2 months for up to a total of 6 doses
  Interventions: Biological: RB-ADSC
- RB-ADSC medium dose (Experimental): Participants will receive 5x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir every 2 months for up to a total of 6 doses
  Interventions: Biological: RB-ADSC
- RB-ADSC high dose (Experimental): Participants will receive 10x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir every 2 months for up to a total of 6 doses
  Interventions: Biological: RB-ADSC

INTERVENTIONS:
Biological: RB-ADSC — Ex Vivo Expanded, Autologous Adipose-Derived Stem Cells (ADSCs)

SUMMARY:
This is a Phase 1b Extension Trial to allow repeat intracerebroventricular injections of RB-ADSCs in subjects previously treated in and successfully completed RBI Protocol RB-ADSC-02. In the previous Phase 1 clinical trial, RB-ADSC-02, subjects with mild to moderate Alzheimer's disease (AD) received a single intraventricular injection of RB-ADSC. RB-ADSC will be delivered intracerebroventricularly every 2 months via the previously implanted Ommaya reservoir for up to 6 injections in total. The primary objective of safety is performed 2 months after the last dose administration at the month 12 follow-up visit. The secondary objective endpoint evaluations of efficacy are performed at the month 6 and 12 visits.

DETAILED DESCRIPTION:
This is a Phase 1b Extension Trial to allow repeat intracerebroventricular injections of RB-ADSCs in subjects previously treated in and successfully completed RBI Protocol RB-ADSC-02. In the previous Phase 1 clinical trial, RB-ADSC-02, subjects with mild to moderate Alzheimer's disease (AD) received a single intraventricular injection of RB-ADSC.

RB-ADSC will be delivered intracerebroventricularly every 2 months via the previously implanted Ommaya reservoir for up to 6 injections in total. Participants will be followed for 2 months after the last administration. The primary objective is safety and tolerability of repeated dosing of RB-ADSC. Adverse events (AEs) and serious adverse events (SAEs) will be assessed by the incidence and severity of dose-limiting toxicity (DLT) and other AEs, incidence and severity of cytokine response syndrome, vital sign measurements, clinical laboratory tests and physical examination. Preliminary efficacy of repeated dosing will be evaluated with clinical assessments (MMSE, FAST, ADAS-Cog), volumetric MRI (NeuroQuant), CSF biomarkers (phosphor-Tau, total-Tau,AB-42), and diagnostic imaging comparison (Amyloid-PET).

ELIGIBILITY:
Inclusion Criteria:

1. Successful completion of the Phase 1 single dose administration study of RB-ADSC, Protocol RB-ADSC-02.
2. Written informed consent to participate in this Phase 1b Extension Study either provided by the participant or a legal representative
3. The participant must have a relative/caregiver who is alert for possible side effects.
4. The caregiver must separately meet the specified inclusion/exclusion criteria for caregivers for this Phase 1b Extension Study.

Exclusion Criteria:

1. Participant experienced treatment related SAE or DLT in Protocol RB-ADSC-02
2. Participants who, in the opinion of the Investigator, are unsuitable for this Phase 1 Extension Study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The safety of repeated RB-ADSC treatment in study participants with AD | up to 12 months
  Safety will be determined by incidence, type and severity of adverse events (AE) and serious adverse events (SAE) graded according to CTCAE v5.0 and CRS revised grading system and defined by clinical relevant findings at every visit and 2 month following last dose in physical examination, vital signs and laboratory data

SECONDARY OUTCOMES:
Change from Baseline in cerebrospinal fluid (CSF) biomarker pTau | Baseline, Month 6, Month 12
  CSF Biomarkers will be measured with the ADmark® phospho-tau/total-tau/ Abeta-42 assay to determine the levels of Phosphorylated-Tau protein in the cerebrospinal fluid (CSF).
Change from Baseline in cerebrospinal fluid (CSF) biomarker Total-Tau | Baseline, Month 6, Month 12
  CSF Biomarkers will be measured with the ADmark® phospho-tau/total-tau/ Abeta-42 assay to determine the levels of Total-Tau protein in the cerebrospinal fluid (CSF).
Change from Baseline in cerebrospinal fluid (CSF) biomarker Ab42 | Baseline, Month 6, Month 12
  CSF Biomarkers will be measured with the ADmark® phospho-tau/total-tau/ Abeta-42 assay to determine the levels of Ab42 in the cerebrospinal fluid (CSF).
Change from Baseline in cerebrospinal fluid (CSF) biomarker ratios reported as amyloid-tau index (ATI) | Baseline, Month 6, Month 12
  CSF Biomarkers will be measured with the ADmark® phospho-tau/total-tau/ Abeta-42 assay to determine the levels of Phosphorylated-Tau protein, Total-Tau protein, and Ab42 in the cerebrospinal fluid (CSF) to calculate ratios and report the amyloid-tau index (ATI).
Change from Baseline in Amyloid Positron Emission Tomography (Amyloid-PET) | Baseline, Month 6, Month 12
  Amyloid-PET will be used to quantitatively assess amyloid plaque deposition in the brain
Change from Baseline in MMSE | Baseline, Month 6, Month 12
  Cognitive function will be evaluated with the Mini Mental State Examination (MMSE). The range for the total MMSE score is 0 to 30, with lower scores indicating greater level of impairment.
Change from Baseline in ADAS-cog13 | Baseline, Month 6, Month 12
  Cognitive function will be assessed using the AD Assessment Scale - Cognitive (ADAS-cog13). The ADAS-Cog13 scale ranges from 0 to 85, with higher scores indicating greater disease severity.
Change from Baseline in FAST | Baseline, Month 6, Month 12
  Functional abilities will be assessed using the Functional Assessment Staging Tool (FAST). The tool consists of seven stages, with higher scores indicating more severe impairment.
Change from Baseline in MoCA | Baseline, Month 6, Month 12
  Mild cognitive impairment and the early onset of dementia will be assessed using the Montreal Cognitive Assessment (MoCA)
Change from Baseline in Volumetric MRI with Contrast | Baseline, Month 6 and Month 12
  Volumetric MRI with contrast of the brain will be used to detect and monitor brain abnormalities.
Change from Baseline in NeuroQuant MRI | Baseline, Month 6 and Month 12
  NeuroQuant MRI will be used to measure volumes of brain structures.

IPD SHARING:
Plan to Share IPD: No